CLINICAL TRIAL: NCT05984082
Title: Checklist for AI in Medical Imaging (CLAIM) Consensus Panel
Acronym: CLAIM
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Charles E. Kahn, Jr., MD, MS, Professor and Vice Chair of Radiology, University of Pennsylvania
Other Study IDs: 853845
Record Dates: First submitted 2023-08-01; First posted 2023-08-09 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Artificial Intelligence; Machine Learning; Diagnostic Imaging
Keywords: Checklist for AI in Medical Imaging (CLAIM); Reporting guideline; Delphi consensus method; Survey

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators will revise the Checklist for AI in Medical Imaging (CLAIM) guideline using Delphi consensus methods. An international panel of physicians, researchers, and journal editors with expertise in AI in medical imaging -- including radiology, pathology, dermatology, GI endoscopy, and ophthalmology -- will complete up to 3 web-based surveys. Participants who complete all survey rounds will be credited as contributors on resulting publications.

DETAILED DESCRIPTION:
The survey will be administered in collaboration with:

* Anthony A. Gatti, PhD (Stanford University)
* Michail E. Klontzas, MD, PhD (University of Crete School of Medicine) *
* Linda Moy, MD (New York University Grossman School of Medicine)
* John Mongan, MD, PhD (University of California San Francisco)
* Seong Ho Park, MD, PhD (University of Ulsan College of Medicine)
* Ali S. Tejani, MD (University of Texas Southwestern Medical School)

(*) Survey administrator

ELIGIBILITY:
Inclusion Criteria:

* More than 70 invited panelists -- physicians, AI researchers, and journal editors -- have agreed to participate in the surveys. Those who participate in all rounds of the survey will be named as contributors in any resulting publications

Exclusion Criteria:

* Non physicians, AI researchers and journal editors

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Physicians, AI researchers and journal editors
Sampling Method: Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Revise the Checklist for AI in Medicine Imaging (CLAIM) guideline | 6 months
  potential revision of the CLAIM guidelines through Delphi consensus process.

CONTACTS AND LOCATIONS:
Overall Officials: Charles E. Kahn, Jr., MD, MS, Principal Investigator — University of Pennsylvania
Locations (1):
- Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Background] Tejani AS, Klontzas ME, Gatti AA, Mongan JT, Moy L, Park SH, Kahn CE Jr; CLAIM 2024 Update Panel. Checklist for Artificial Intelligence in Medical Imaging (CLAIM): 2024 Update. Radiol Artif Intell. 2024 Jul;6(4):e240300. doi: 10.1148/ryai.240300. PMID 38809149